CLINICAL TRIAL: NCT01134003
Title: A Large Multi-Center Database of Women Who Have Had and Are Going to Have Surgical Correction of Their Pelvic Organ Prolapse Using the Gynecare Prolift System
Status: Completed | Type: Observational
Sponsor: The Institute of Pelvic Medicine & Reconstructive Surgery, Allentown, Pennsylvania (Other)
Responsible Party: Dr. Vincent Lucente, Institute for Female Pelvic Medicine
Other Study IDs: SLHN 2007-98
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Last update posted 2010-05-31 (Estimated); Status verified 2010-05

CONDITIONS: Pelvic Organ Prolapse
Keywords: Gynecare Prolift; Pelvic organ prolapse; forming a large database of women who have recieve Gynecare prolift system
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
retrospective and prospective data collection for a database. Patients will have had or are going to have a repair of their pelvic organ prolapse using the Gynecare mesh Prolift System

ELIGIBILITY:
Inclusion Criteria:

* women recieving surgery for their pelvic organ prolapse using the Gynecare mesh kit called Prolift

Exclusion Criteria:

* none

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: women receiving surgery for their pelvic organ prolapse using the Gynecare mesh kit called Prolift
Sampling Method: Probability Sample
Dates: Start 2008-01; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Female Pelvic Medicine and Reconstructive Surgery, Allentown, Pennsylvania, United States